CLINICAL TRIAL: NCT06928935
Title: Digital Dialectical Behavioural Therapy (d-DBT) for Youth at Clinical High Risk (CHR) for Psychosis: An Exploratory Multi-Methods Study
Brief Title: Digital Dialectical Behavioural Therapy (d-DBT) for Youth at Clinical High Risk (CHR) for Psychosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Omair Husain, Clinician Scientist, Psychiatrist, Associate Professor, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/007
Record Dates: First submitted 2025-03-26; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Clinical High Risk for Psychosis (CHR)
Keywords: digital therapy; dialectical behavioural therapy; emotional dysregulation; mental health intervention; digital mental health; clinical high risk for psychosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be conducted by a blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): This arm will receive the d-DBT intervention.
  Interventions: Behavioral: d-DBT
- Control (Treatment as Usual) (No Intervention): This arm will not receive the intervention. Participants continue with standard outpatient care, including routine healthcare provider appointments and medication management.

INTERVENTIONS:
Behavioral: d-DBT — d-DBT is an 8-week self-led online intervention that teaches mindfulness, emotional regulation, distress tolerance, and interpersonal effectiveness skills. Participants receive weekly digital navigator check-ins.
  Arms: Experimental

SUMMARY:
This study examines the feasibility and acceptability of a digital dialectical behavior therapy (d-DBT) intervention for youth at clinical high risk (CHR) for psychosis. The study aims to assess the acceptability of the intervention to the CHR population, the feasibility of conducting a larger-scale clinical efficacy trial and the potential benefits in improving emotional regulation, reducing psychiatric symptoms, and enhancing overall functioning. Participants will be randomized to receive either the d-DBT intervention or treatment as usual over eight weeks.

DETAILED DESCRIPTION:
This study evaluates the feasibility, acceptability, and preliminary efficacy of digital Dialectical Behavior Therapy (d-DBT) for youth at Clinical High Risk (CHR) for psychosis. Given the limited availability of evidence-based digital interventions tailored to this group, this trial explores whether a digital DBT approach can address emotion dysregulation, mood symptoms, and functional impairments, which are common in CHR populations and may contribute to distress and progression of disease.

Participants will be randomized to receive either d-DBT or treatment-as-usual (TAU). The intervention is designed to be self-directed, incorporating, interactive exercises, and skill-building modules targeting emotional regulation, distress tolerance, mindfulness, and substance use. Primary outcomes include measuring feasibility, acceptability, and usability. Secondary measures will evaluate preliminary clinical outcomes related to psychiatric symptoms, substance use, and functioning. Results will inform future adaptations, larger trials, and clinical applications.

ELIGIBILITY:
Inclusion Criteria:

1. Be 16-29 years old.
2. Being competent and willing to consent to study participation.
3. Meets CHR criteria for a psychosis risk syndrome based on the Structured Interview for Psychosis Risk Syndromes (SIPS) within the past 3 years.

Exclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of psychotic disorder (e.g., schizophrenia spectrum disorder, mood disorder with psychotic features)
2. Diagnosis of intellectual disability
3. Severe developmental disorder
4. Acute suicidality requiring immediate life-saving intervention (i.e., inpatient psychiatric care).
5. Receiving any additional psychotherapy interventions or structured digital mental health support during the study period.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 8 weeks
  The percentage of participants enrolled in the study, with higher numbers indicating greater recruitment success.
Retention | 8 weeks
  The percentage of participants who remain enrolled by the end of the study, with higher numbers indicating better retention.
Adherence | 8 weeks
  Percentage of modules completed; higher percentages indicate greater adherence.
Client Satisfaction Questionnaire | 8 weeks
  A Likert scale from 1-4, total scores range from 8-32, with higher scores indicating greater satisfaction.
System Usability Scale | 8 weeks
  A 10-item Likert scale scored from 1-5; total scores range from 0-100, with higher scores indicating greater perceived usability.

SECONDARY OUTCOMES:
Structured Interview for Psychosis-risk Syndromes (SIPS) | Baseline and 8 weeks
  The Structured Interview for Prodromal Symptoms (SIPS) is a widely used structured interview for diagnosing a CHR syndrome for psychosis and cases of first episode psychosis. It contains a severity rating scale (the Scale Of Psychosis-risk Symptoms, or SOPS). It is a 6-point scale, with higher scores indicating higher severity.
PRIME-Revised (PRIME-R) | Baseline and 8 weeks
  A 12-item Likert scale (0-6) measuring severity of prodromal psychotic symptoms; total scores range from 0-72, with higher scores indicating greater symptom severity.
Borderline Symptom List (BSL-23) | Baseline and 8 weeks
  A 23-item Likert scale scored from 0-4; total scores range from 0-92, with higher scores indicating greater severity of borderline personality symptoms.
Brief Difficulties in Emotion Regulation Scale (DERS-16) | Baseline and 8 weeks
  A 16-item Likert scale scored from 1-5; total scores range from 16-80, with higher scores indicating greater difficulties in emotion regulation.
State-Trait Anxiety Inventory (STAI) | Baseline and 8 weeks
  A 40-item measure (20 items for state anxiety, 20 items for trait anxiety) scored on a 4-point Likert scale (1-4); total scores range from 20-80 per subscale, with higher scores indicating greater anxiety.
Calgary Depression Scale for Schizophrenia (CDSS) | Baseline and 8 weeks
  A 9-item clinician-rated scale scored from 0-3 per item; total scores range from 0-27, with higher scores indicating greater depressive symptom severity.
Global Functioning: Social and Role Scales | Baseline and 8 weeks
  Two clinician-rated scales ranging from 1-10 each, assessing social and role functioning; higher scores indicate better overall functioning.
Connor-Davidson Resilience Scale (CD-RISC) | Baseline and 8 weeks
  A 25-item Likert scale scored from 0-4; total scores range from 0-100, with higher scores indicating greater resilience.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline and 8 weeks
  A structured clinical interview assessing suicidal ideation and behavior severity; scores include ideation severity (0-5) and behavior presence; higher scores indicate greater suicide risk.
MATRICS Consensus Cognitive Battery (MCCB) | Baseline and 8 weeks
  A standardized cognitive assessment comprising 10 tests across 7 domains; total composite T-scores typically range from 10-90, with higher scores indicating better cognitive functioning.
Timeline Follow Back (TLFB) | Baseline and 8 weeks
  A calendar-based assessment method recording daily cannabis, alcohol, and tobacco use over the past 7 days; higher frequency or quantity indicates greater substance use.
Cannabis Use Disorders Identification Test-Revised (CUDIT-R) | Baseline and 8 weeks
  An 8-item screening tool scored from 0-32; higher scores indicate increased risk or severity of cannabis use disorder.
Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory (DFAQ-CU) | Baseline and 8 weeks
  A self-report questionnaire assessing detailed patterns of cannabis use, including daily sessions, frequency, age of first use, and quantity consumed; higher values indicate greater cannabis involvement.
Adolescent Alcohol and Drug Involvement Scale (AADIS) | Baseline and 8 weeks
  A brief screening tool scoring substance use involvement from 0-79; higher scores indicate greater severity of alcohol and drug involvement.

CONTACTS AND LOCATIONS:
Overall Officials: M. Omair Husain, MBBS, MRCPsych, Principal Investigator — The Centre for Addiction and Mental Health (CAMH)
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available on reasonable request from the principal investigator.

REFERENCES:
- [Background] Lawlor C, Vitoratou S, Hepworth C, Jolley S. Self-reported emotion regulation difficulties in psychosis: Psychometric properties of the Difficulties in Emotion Regulation Scale (DERS-16). J Clin Psychol. 2021 Oct;77(10):2323-2340. doi: 10.1002/jclp.23164. Epub 2021 May 10. PMID 33971018
- [Background] Adamson SJ, Kay-Lambkin FJ, Baker AL, Lewin TJ, Thornton L, Kelly BJ, Sellman JD. An improved brief measure of cannabis misuse: the Cannabis Use Disorders Identification Test-Revised (CUDIT-R). Drug Alcohol Depend. 2010 Jul 1;110(1-2):137-43. doi: 10.1016/j.drugalcdep.2010.02.017. Epub 2010 Mar 26. PMID 20347232
- [Background] Robinson SM, Sobell LC, Sobell MB, Leo GI. Reliability of the Timeline Followback for cocaine, cannabis, and cigarette use. Psychol Addict Behav. 2014 Mar;28(1):154-62. doi: 10.1037/a0030992. Epub 2012 Dec 31. PMID 23276315
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Miller TJ, McGlashan TH, Rosen JL, Cadenhead K, Cannon T, Ventura J, McFarlane W, Perkins DO, Pearlson GD, Woods SW. Prodromal assessment with the structured interview for prodromal syndromes and the scale of prodromal symptoms: predictive validity, interrater reliability, and training to reliability. Schizophr Bull. 2003;29(4):703-15. doi: 10.1093/oxfordjournals.schbul.a007040. PMID 14989408
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Neacsiu AD, Eberle JW, Kramer R, Wiesmann T, Linehan MM. Dialectical behavior therapy skills for transdiagnostic emotion dysregulation: a pilot randomized controlled trial. Behav Res Ther. 2014 Aug;59:40-51. doi: 10.1016/j.brat.2014.05.005. Epub 2014 May 27. PMID 24974307
- [Background] Linehan MM, Korslund KE, Harned MS, Gallop RJ, Lungu A, Neacsiu AD, McDavid J, Comtois KA, Murray-Gregory AM. Dialectical behavior therapy for high suicide risk in individuals with borderline personality disorder: a randomized clinical trial and component analysis. JAMA Psychiatry. 2015 May;72(5):475-82. doi: 10.1001/jamapsychiatry.2014.3039. PMID 25806661
- [Background] Woods SW, Addington J, Cadenhead KS, Cannon TD, Cornblatt BA, Heinssen R, Perkins DO, Seidman LJ, Tsuang MT, Walker EF, McGlashan TH. Validity of the prodromal risk syndrome for first psychosis: findings from the North American Prodrome Longitudinal Study. Schizophr Bull. 2009 Sep;35(5):894-908. doi: 10.1093/schbul/sbp027. Epub 2009 Apr 21. PMID 19386578
- [Background] Addington J, van der Gaag M. Psychosocial treatments for clinical high risk individuals. Schizophr Bull. 2015 Jan;41(1):22. doi: 10.1093/schbul/sbu140. Epub 2014 Oct 14. No abstract available. PMID 25316912
- [Background] Fusar-Poli P, De Micheli A, Signorini L, Baldwin H, Salazar de Pablo G, McGuire P. Real-world long-term outcomes in individuals at clinical risk for psychosis: The case for extending duration of care. EClinicalMedicine. 2020 Oct 7;28:100578. doi: 10.1016/j.eclinm.2020.100578. eCollection 2020 Nov. PMID 33294806
- [Derived] Hedemann TL, Lu Y, Campitelli S, Hawke LD, Shen N, Saperia S, Jones BDM, Strudwick G, Wilks CR, Wang W, Solmi M, Grossman M, Husain MI, Kozloff N, Foussias G, Husain MO. Adaptation and evaluation of a digital dialectical behaviour therapy for youth at clinical high risk for psychosis: A protocol for a feasibility randomized controlled trial. PLoS One. 2025 Dec 23;20(12):e0339163. doi: 10.1371/journal.pone.0339163. eCollection 2025. PMID 41433354